CLINICAL TRIAL: NCT05089656
Title: A Randomized, Sham-controlled, Double-blind Study to Evaluate the Efficacy and Safety of Intrathecal OAV101 in Type 2 Spinal Muscular Atrophy (SMA) Patients Who Are ≥ 2 to < 18 Years of Age, Treatment Naive, Sitting, and Never Ambulatory
Brief Title: Efficacy and Safety of Intrathecal OAV101 (AVXS-101) in Pediatric Patients With Type 2 Spinal Muscular Atrophy (SMA)
Acronym: STEER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COAV101B12301; 2021-003474-31 (EudraCT Number)
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Results first posted 2025-12-08 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Spinal Muscular Atrophy
Keywords: Zolgensma; OAV101; AVXS 101; gene therapy; Muscle atrophy; SMA; spinal muscular atrophy; muscle function; myopathy; muscle wasting; atrophied muscle; loss of muscle strength; pediatric
MeSH Terms: conditions — Spinal Muscular Atrophies of Childhood; Muscular Atrophy; Muscular Atrophy, Spinal; Muscular Diseases | interventions — Zolgensma

STUDY DESIGN:
Intervention Model Description: A participant will receive a single, one-time dose of OAV101.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OAV101 in Treatment Period 1; Sham Control in Treatment Period 2 (Experimental): OAV101 administered as a single, one-time intrathecal dose of 1.2 x 10^14 vector genomes (vg) in Treatment Period 1; Sham Control in Treatment Period 2 (Week 52 +1 day).
  Interventions: Genetic: OAV101
- Sham control in Treatment Period 1; OAV101 in Treatment Period 2 (Sham Comparator): A skin prick in the lumbar region in Treat Period 1; OAV101 administered as a single, one-time intrathecal dose of 1.2 x 10^14 vector genomes (vg) in Treatment Period 2 (Week 52 +1 day)
  Interventions: Procedure: Sham control

INTERVENTIONS:
Genetic: OAV101 — Gene therapy
  Other Names: Zolgensma; AVXS-101
  Arms: OAV101 in Treatment Period 1; Sham Control in Treatment Period 2
Procedure: Sham control — The sham procedure will consist of a small needle prick on the lower back at the location where the LP injection is normally made. The needle will break the skin, but no needle insertion for lumbar puncture will occur.
  Arms: Sham control in Treatment Period 1; OAV101 in Treatment Period 2

SUMMARY:
This was a Phase III multi-center, single dose (1.2 x 10^14 vector genomes), randomized, sham controlled, double-blind study that investigates the efficacy, safety and tolerability of OAV101B in treatment naive, sitting and never ambulatory SMA patients 2 to <18 years of age.

DETAILED DESCRIPTION:
Eligible participants received a single administration of OAV101B at the dose of 1.2 x 10^14 vector genomes intrathecally or the sham procedure on Day 1 (Treatment Period 1), and were followed for a period of 52 weeks for Period 1. In Period 2, participants who received the sham treatment in Period 1 were administered OAV101B, and participants who received OAV101B in Period 1 underwent the sham procedure. Participants were followed up for 12 weeks in Period 2.

The study consisted of a Screening and Baseline Period followed by two Treatment and Follow-up Periods. Participants were admitted to the hospital on Day 1 (or Day -1 as per local standards of care). After receiving OAV101B or the sham procedure on Day 1, participants underwent in-patient safety monitoring through Day 2 and optionally for Day 3.

After Period 1, eligible participants could continue to Period 2 subsequently entering Period 2 in a rolling seamless fashion as participants completed Follow-up Period 1. In Treatment Period 2, eligible participants who received a sham procedure on Study Day 1 of Treatment Period 1 were hospitalized to receive OAV101B on Week 52 + 1 day and participants who received OAV101B on Study Day 1 of Treatment Period 1 were hospitalized to receive a sham procedure on the Week 52 + 1 Day. The total duration of the study including both Period 1 and Period 2 was 64 weeks. At the end of the study, all participants who received OAV101B were eligible to enroll in a long-term follow-up study to monitor long-term safety and efficacy.

Approximately 125 participants were planned to be randomized in a 3:2 ratio to receive OAV101B (N= ~75) or a sham procedure (N= ~50). The unequal randomization ratio allowed more participants to receive active treatment in Period 1. It was anticipated that approximately 65 randomized participants would be aged 2 to <5 years and approximately 60 randomized participants would be aged 5 to <18 years.

ELIGIBILITY:
Key Inclusion criteria:

* Diagnostic confirmation during screening period of 5q SMA
* The patient must be treatment naive (historical or current use) for all SMN-targeting therapies (e.g., risdiplam (Evrysdi) and nusinersen (Spinraza)).
* Onset of clinical signs and symptoms at ≥ 6 months of age
* A complete Hammersmith Functional Motor Scale - Expanded (HFMSE) assessment during the screening period for trial eligibility
* Able to sit independently at screening, but has never had the ability to walk independently.

Key Exclusion criteria:

* Anti-adeno-associated virus serotype 9 (AAV9) antibody titer reported as elevated (reference to > 1:50 or validated result consistent with being elevated) at screening as determined by sponsor designated lab.
* Infectious process (e.g., viral, bacterial) or febrile illness within 30 days prior to OAV101 treatment or sham procedure
* Hepatic dysfunction (i.e. alanine aminotransferase (ALT), total bilirubin, gamma-glutamyl transferase (GGT) or glutamate dehydrogenase (GLDH), > upper limit of normal (ULN).
* Requiring invasive ventilation, awake noninvasive ventilation for > 6 hours during a 24-hour period, noninvasive ventilation for > 12 hours during a 24-hour period or requiring tracheostomy
* Complications at screening that would interfere with motor efficacy assessments including but not limited to, severe contractures or Cobb angle > 40 in a sitting position
* Surgery for scoliosis or hip fixation in the 12 months prior to Screening or planned within the next 64 weeks
* Clinically significant sensory abnormalities in the neurological examination at Screening

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 126 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2025-04-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (6):
  - Connecticut Children's Medical Center, Farmington, Connecticut
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Clinic for Special Children, Strasburg, Pennsylvania
  - St Jude Children's Research Hospital, Memphis, Tennessee
  - Child Hosp Of The Kings Daughters, Norfolk, Virginia
  - Children's Specialty Group/CHKD, Norfolk, Virginia
- Brazil (2):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, São Paulo, São Paulo
- China (8):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Novartis Investigative Site, Beijing
- Denmark (2):
  - Novartis Investigative Site, Copenhagen
  - Paediatric Neurology, Copenhagen
- India (7):
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - AIIMS, Ansari Nagar, New Delhi, New Delhi
  - Novartis Investigative Site, Kolkata, West Bengal
  - Novartis Investigative Site, Hyderabad
  - Novartis Investigative Site, Mumbai
  - P.D. Hinduja National Hospital & MRC, Mumbai
- Novartis Investigative Site, Kuala Lumpur, Malaysia
- Mexico (3):
  - Hospital Civil De Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City, Mexico City
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- South Africa (2):
  - Novartis Investigative Site, Cape Town
  - Red Cross War Memorial Childrens Hospital, Cape Town
- Taiwan (2):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Novartis Investigative Site, Kaohsiung City
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Siriraj Hospital, Bangkok
- Vietnam (2):
  - National Children's Hospital, Hanoi
  - Novartis Investigative Site, Hanoi

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on https://www.clinicalstudydatarequest.com/.
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Proud CM, Vu DC, Wilmshurst JM, Sanmaneechai O, Gulati S, Xiong H, Moreno HC, Tay SKH, Thong MK, Born AP, Banzzatto Ortega A, Jong YJ, Al-Muhaizea MA, Lee AW, Visootsak J, Tauscher-Wisniewski S, Alecu I, Parlikar R, Finkel RS; STEER Study Group. Intrathecal onasemnogene abeparvovec in treatment-naive patients with spinal muscular atrophy: a phase 3, randomized controlled trial. Nat Med. 2025 Dec 8. doi: 10.1038/s41591-025-04103-w. Online ahead of print. PMID 41360993
- See also: Results for COAV101B12301 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18373
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2997
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=806

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 121 total participants were treated with a single dose of OAV101B (either in Period 1 (even if they did not complete Period 1) or Period 2).
Groups:
- OAV101 First, Then Sham Control: OAV101 administered as a single, one-time intrathecal dose of 1.2 x 10^14 vector genomes (vg) in Period 1, then a skin prick in the lumbar region without any medication in Period 2
- Sham Control First, Then OAV101: A skin prick in the lumbar region without any medication in Period 1, then OAV101 administered as a single, one-time intrathecal dose of 1.2 x 10^14 vector genomes (vg) in Period 2
Period: Period 1 - First Intervention (52 weeks)
Arm/Group | OAV101 First, Then Sham Control | Sham Control First, Then OAV101
Started | 75 | 51
Patients completed follow-up period 1 | 73 | 50
Patients completed follow-up period 1 but did not enter treatment period 2 | 6 | 4
Patient who completed Week 48 but not Week 52 | 1 | 0
Primary reason for not entering treatment period 2 (Protocol-specified withdrawal criterion met) | 6 | 4
Completed (Patients completed follow-up period 1 and entered treatment period 2) | 67 | 46
Not Completed | 8 | 5
Not completed — Physician Decision | 1 | 0
Not completed — Guardian decision | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Protocol-specified withdrawal criterion met | 6 | 4
Period: Period 2 - 2nd Intervention (12 weeks)
Arm/Group | OAV101 First, Then Sham Control | Sham Control First, Then OAV101
Started | 67 | 46
Completed | 67 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OAV101 First, Then Sham Control | Sham Control First, Then OAV101 | Total
Number analyzed (Participants) | 75 | 51 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.71 (3.575) | 5.68 (3.045) | 5.70 (3.358)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 23 | 64
  Male | 34 | 28 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 5 | 7
  Asian | 49 | 25 | 74
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 4 | 9
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline at the End of Period 1 in the Hammersmith Functional Motor Scale Expanded - Total Score - in the ≥ 2 to < 18 Years Age Group
Description: The HFMSE is a validated SMA specific assessment devised for use in children with SMA to give objective information on motor ability and clinical progression. The HFMSE contains 33 items rated from 0 (unable to perform) to 2 (performs without modification/adaptation/compensation). Total scores range from 0-66. Higher scores indicate higher levels of motor ability.
Time Frame: Baseline, Week 52 (or Week 48)
Population: Full Analysis Set - all participants who were treated in treatment period 1 with a valid measurement (including 1 pt who dropped out between Week 48 and week 52; The data collected at Week 48 are included in this table.) (Participants who early terminated before Week 48 are not included).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | OAV101 First, Then Sham Control | Sham Control First, Then OAV101
Number analyzed (Participants) | 74 | 50
Scores on a scale | 2.39 (0.439) | 0.51 (0.532)
Statistical Analysis 1: Comparison: OAV101 First, Then Sham Control vs Sham Control First, Then OAV101; Change from baseline at End of Follow-up Period 1; Test type: Superiority; p = 0.0074, Mixed Models Analysis; LS-Means difference = 1.88, 95% CI 2-sided [0.51 to 3.25], Standard Error of Mean 0.690

2. Secondary Outcome: Change From Baseline in HFMSE Total Score at the End of Follow-up Period 1 in Treated Patients Compared to Sham Controls in the ≥ 2 to < 5 Years Age Group
Description: as for outcome 1
Time Frame: Baseline, Week 52 (or Week 48)
Population: Full Analysis Set - all participants who were treated in treatment period 1 with a valid measurement in the 2 to <5 years age group. (Participants who early terminated before Week 48 are not included.)
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | OAV101 First, Then Sham Control | Sham Control First, Then OAV101
Number analyzed (Participants) | 41 | 29
Scores on a scale | 3.00 (0.569) | 1.56 (0.683)
Statistical Analysis 1: Comparison: OAV101 First, Then Sham Control vs Sham Control First, Then OAV101; Change from baseline at End of Follow-up Period 1; Test type: Superiority; p = 0.1097, Mixed Models Analysis; LS-Means - difference = 1.44, 95% CI 2-sided [-0.33 to 3.22], Standard Error of Mean 0.889

3. Secondary Outcome: Change From Baseline in Revised Upper Limb Module (RULM) Total Score at the End of Follow-up Period 1 in Treated Patients Compared to Sham Controls in the ≥ 2 to < 18 Years Age Group
Description: The RULM is a validated SMA specific assessment of motor performance in the upper limbs from childhood through adulthood in ambulatory and non-ambulatory individuals with SMA. The scale consists of 19 scorable items: 18 items scored on 0 (unable) to 2 (full achievement) scale, and one item that is scored from 0 (unable) to 1 (able). Total scores range from 0-37 points. Higher scores reflect higher level of motor ability.
Time Frame: Baseline, Week 52 (or Week 48)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | OAV101 First, Then Sham Control | Sham Control First, Then OAV101
Number analyzed (Participants) | 74 | 50
Scores on a scale | 2.44 (0.381) | 0.92 (0.462)
Statistical Analysis 1: Comparison: OAV101 First, Then Sham Control vs Sham Control First, Then OAV101; Change from baseline at End of Follow-up Period 1; Test type: Superiority; p = 0.0122, Mixed Models Analysis; LS-Means difference = 1.52, 95% CI 2-sided [0.34 to 2.71], Standard Error of Mean 0.599

4. Secondary Outcome: Change From Baseline in the RULM Total Score at the End of Follow-up Period 1 in Treated Patients Compared to Sham Controls in the ≥ 2 to < 5 Years Age Group
Description: The RULM is a validated SMA specific assessment of motor performance in the upper limbs from childhood through adulthood in ambulatory and non-ambulatory individuals with SMA. The scale consists of 19 scorable items: 18 items scored on a 0 (unable) to 2 (full achievement) scale, and one item that is scored from 0 (unable) to 1 (able). Total scores range from 0-37 points. Higher scores reflect higher level of motor ability.
Time Frame: Baseline, Week 52 (or Week 48)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | OAV101 First, Then Sham Control | Sham Control First, Then OAV101
Number analyzed (Participants) | 41 | 29
Scores on a scale | 3.27 (0.535) | 1.82 (0.642)
Statistical Analysis 1: Comparison: OAV101 First, Then Sham Control vs Sham Control First, Then OAV101; Change from baseline at End of Follow-up Period 1; Test type: Superiority; p = 0.0873, Mixed Models Analysis; LS-Means difference = 1.45, 95% CI 2-sided [-0.22 to 3.12], Standard Error of Mean 0.836

5. Secondary Outcome: % of Participants Who Achieved at Least a 3-point Improvement From Baseline in HFMSE Total Score at the End of Follow-up Period 1 in the ≥ 2 to < 18 Years Age Group
Description: as for outcome 1
Time Frame: Baseline, Week 52 (or Week 48) (end of Period 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | OAV101 First, Then Sham Control | Sham Control First, Then OAV101
Number analyzed (Participants) | 74 | 50
% of participants | 39.2 [28.07 to 50.31] | 26.0 [13.84 to 38.16]
Statistical Analysis 1: Comparison: OAV101 First, Then Sham Control vs Sham Control First, Then OAV101; End of Followup Period 1 (Week 52); Test type: Superiority; p = 0.0879, Regression, Logistic; Odds Ratio (OR) = 2.03, 95% CI 2-sided [0.90 to 4.57]

6. Secondary Outcome: % of Participants Who Achieved at Least a 3-point Improvement From Baseline in HFMSE Total Score at the End of Follow-up Period 1 for Participants Aged ≥ 2 to < 5 Years
Description: as for outcome 1
Time Frame: Baseline, Week 52 (or Week 48)(end of Period 1)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | OAV101 First, Then Sham Control | Sham Control First, Then OAV101
Number analyzed (Participants) | 41 | 29
% of participants | 48.8 [33.48 to 64.08] | 37.9 [20.27 to 55.59]
Statistical Analysis 1: Comparison: OAV101 First, Then Sham Control vs Sham Control First, Then OAV101; End of Followup Period 1 (Week 52); Test type: Superiority; p = 0.6448, Regression, Logistic; Odds Ratio (OR) = 1.27, 95% CI 2-sided [0.46 to 3.56]

7. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
  A Treatment Emergent Adverse Event (TEAE) is defined as an event that emerges during treatment, having been absent pretreatment, or worsens relative to the pretreatment state.
  The occurrence of AEs must be sought by non-directive questioning of the participant at each visit during the study. Adverse events also may be detected when they are volunteered by the participant during or between visits or through physical examination findings, laboratory test findings, or other assessments.
  pt = participant pts = participants
Time Frame: Adverse events are reported from the start of treatment period 1 plus 64 weeks, up to a maximum time period of 64 weeks.
Population: Safety analysis set - all treated pts.
  AEs for Periods 1 and 2 are combined in the overall OAV101 arm because the same active treatment (and same single dose) was administered in either Period1 or 2. Because this is a gene therapy, which permanently impacts the genetics of the study pt, pts randomized to OAV101 in Period 1 are still considered on treatment with OAV101 in Period 2 (after receiving sham control in Period 2). Therefore, AEs for the Sham arm can only be considered from Period 1.
Measure: Count of Participants; unit: Participants
Groups:
- OAV101 Period 1: OAV101 administered as a single, one-time intrathecal dose of 1.2 x 10^14 vector genomes (vg) in Period 1
- Sham Control Period 1: A skin prick in the lumbar region without any medication in Period 1
- Overall OAV101 in Periods 1 and 2: OAV101 administered as a single, one-time intrathecal dose of 1.2 x 10^14 vector genomes (vg).
  * For participants randomized to OAV101B in Period 1: All AEs from Period 1 and 2
  * For participants randomized to the sham control in Period 1 and who were administered OAV101 in Period 2: All AEs from Period 2
Arm/Group | OAV101 Period 1 | Sham Control Period 1 | Overall OAV101 in Periods 1 and 2
Number analyzed (Participants) | 75 | 51 | 121
Participants
  Any treatment-emergent adverse event | 74 | 46 | 104
  Any treatment-emergent adverse event related to study treatment | 27 | 5 | 36
  Any serious treatment-emergent adverse event | 21 | 17 | 34
  Any serious treatment-emergent adverse event related to study treatment | 8 | 1 | 12
  Any severe treatment-emergent adverse event | 8 | 9 | 12
  Any treatment-emergent adverse event leading to study discontinuation | 0 | 1 | 0
  Any treatment-emergent adverse event leading to death | 0 | 0 | 0
  Any treatment-emergent adverse event of special interest | 12 | 7 | 21

8. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI)
Description: An AESI is primarily defined by using standard Medical Dictionary for Regulatory Activities (MedDRA) queries, and identified as follows:
  * Hepatotoxicity
  * Thrombocytopenia
  * Cardiac adverse events
  * Signs and symptoms that may be suggestive of dorsal root ganglia toxicity
  * Thrombotic microangiopathy
  * New malignancies
  Adverse events for Periods 1 and 2 are combined in the overall OAV101 arm because the same active treatment (and same single dose) was administered in either Period1 or Period 2. Because this is a gene therapy, which permanently impacts the genetics of the study participant, participants randomized to OAV101 in Period 1 are still considered on treatment with OAV101 in Period 2 (after receiving sham control in Period 2). Therefore, adverse events for the Sham arm can only be considered from Period 1.
Time Frame: Adverse events are reported from the start of treatment period 1 plus 64 weeks, up to a maximum time period of 64 weeks.
Population: Safety analysis set - all treated participants.
Measure: Count of Participants; unit: Participants
Arm/Group | OAV101 Period 1 | Sham Control Period 1 | Overall OAV101 in Periods 1 and 2
Number analyzed (Participants) | 75 | 51 | 121
Participants
  Hepatotoxicity | 7 | 5 | 10
  Transient thrombocytopenia | 4 | 2 | 9
  Cardiac adverse events | 0 | 0 | 0
  Signs and symptoms that may be suggestive of dorsal root ganglia toxicity | 2 | 1 | 3
  Thrombotic microangiopathy | 0 | 0 | 0
  New malignancies | 0 | 0 | 0

9. Secondary Outcome: Number (and Percentage) of Patients With Intracardiac Thrombi
Description: Intracardiac thrombi is defined as the presence of thrombus on post-baseline echocardiograms.
  Events for Periods 1 and 2 are combined in the overall OAV101 arm because the same active treatment (and same single dose) was administered in either Period1 or Period 2. Because this is a gene therapy, which permanently impacts the genetics of the study participant, participants randomized to OAV101 in Period 1 are still considered on treatment with OAV101 in Period 2 (after receiving sham control in Period 2). Therefore, events for the Sham arm can only be considered from Period 1.
Time Frame: Baseline up to 64 weeks
Population: Safety analysis set - all treated participants.
Measure: Count of Participants; unit: Participants
Groups:
- Overall OAV101 in Periods 1 and 2: OAV101 administered as a single, one-time intrathecal dose of 1.2 x 10^14 vector genomes (vg).
  * For participants randomized to OAV101B in Period 1: All intracardiac thrombi events from Period 1 and 2
  * For participants randomized to the sham control in Period 1 and who were administered OAV101 in Period 2: All intracardiac thrombi events from Period 2
Arm/Group | OAV101 Period 1 | Sham Control Period 1 | Overall OAV101 in Periods 1 and 2
Number analyzed (Participants) | 75 | 51 | 121
Participants | 0 | 1 | 1

10. Secondary Outcome: Number(and Percentage) of Patients With Low Cardiac Function
Description: Low cardiac function is defined as left ventricular ejection fraction <56% or left ventricular fractional shortening <28% on post-baseline echocardigrams.
  Events for Periods 1 and 2 are combined in the overall OAV101 arm because the same active treatment (and same single dose) was administered in either Period1 or Period 2. Because this is a gene therapy, which permanently impacts the genetics of the study participant, participants randomized to OAV101 in Period 1 are still considered on treatment with OAV101 in Period 2 (after receiving sham control in Period 2). Therefore, events for the Sham arm can only be considered from Period 1.
Time Frame: Baseline up to 64 weeks
Population: Safety analysis set - all treated participants.
Measure: Count of Participants; unit: Participants
Groups:
- Overall OAV101 in Periods 1 and 2: OAV101 administered as a single, one-time intrathecal dose of 1.2 x 10^14 vector genomes (vg).
  * For participants randomized to OAV101B in Period 1: All low cardiac function events from Period 1 and 2
  * For participants randomized to the sham control in Period 1 and who were administered OAV101 in Period 2: All low cardiac function events from Period 2
Arm/Group | OAV101 Period 1 | Sham Control Period 1 | Overall OAV101 in Periods 1 and 2
Number analyzed (Participants) | 75 | 51 | 121
Participants | 8 | 9 | 17

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are reported from the start of treatment period 1 plus 64 weeks, up to a maximum time period of 64 weeks.
Description: AEs for Periods 1 and 2 are combined in the overall OAV101 arm because the same active treatment (and same single dose) was administered in either Period1 or Period 2. Because this is a gene therapy, which permanently impacts the genetics of the study participant, participants randomized to OAV101 in Period 1 are still considered on treatment with OAV101 in Period 2 (after receiving sham control in Period 2). Therefore, AEs for the Sham arm can only be considered from Period 1.
Groups:
- Overall OAV101 in Periods 1 and 2: OAV101 administered as a single, one-time intrathecal dose of 1.2 x 10^14 vector genomes (vg). -For participants randomized to OAV101B in Period 1: All AEs from Period 1 and 2 -For participants randomized to the sham control in Period 1 and who were administered OAV101 in Period 2: All AEs from Period 2
Arm/Group | OAV101 Period 1 | Sham Control Period 1 | Overall OAV101 in Periods 1 and 2
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/51 | 0/121
Serious Adverse Events (participants affected / at risk) | 21/75 | 17/51 | 34/121
Other Adverse Events (participants affected / at risk) | 63/75 | 43/51 | 85/121
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OAV101 Period 1 (N=75) | Sham Control Period 1 (N=51) | Overall OAV101 in Periods 1 and 2 (N=121)
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 5
Pyrexia (General disorders and administration site conditions) | 1 | 0 | 3
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 1
Coronavirus pneumonia (Infections and infestations) | 1 | 0 | 1
Hand-foot-and-mouth disease (Infections and infestations) | 0 | 1 | 0
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 0 | 2
Lower respiratory tract infection (Infections and infestations) | 2 | 4 | 2
Metapneumovirus infection (Infections and infestations) | 1 | 0 | 1
Mycoplasma infection (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 9 | 7 | 16
Pneumonia aspiration (Infections and infestations) | 0 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 2 | 1
Pneumonia mycoplasmal (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 2 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OAV101 Period 1 (N=75) | Sham Control Period 1 (N=51) | Overall OAV101 in Periods 1 and 2 (N=121)
Constipation (Gastrointestinal disorders) | 11 | 11 | 15
Diarrhoea (Gastrointestinal disorders) | 1 | 8 | 2
Nausea (Gastrointestinal disorders) | 4 | 3 | 6
Vomiting (Gastrointestinal disorders) | 13 | 6 | 18
Pyrexia (General disorders and administration site conditions) | 19 | 12 | 23
Bronchitis (Infections and infestations) | 4 | 3 | 7
Influenza (Infections and infestations) | 4 | 5 | 5
Lower respiratory tract infection (Infections and infestations) | 6 | 4 | 7
Nasopharyngitis (Infections and infestations) | 8 | 5 | 11
Pharyngitis (Infections and infestations) | 3 | 4 | 5
Pneumonia (Infections and infestations) | 0 | 3 | 1
Respiratory tract infection (Infections and infestations) | 3 | 3 | 5
Upper respiratory tract infection (Infections and infestations) | 26 | 15 | 34
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Dizziness (Nervous system disorders) | 4 | 1 | 5
Headache (Nervous system disorders) | 7 | 2 | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 15
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 8
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 2
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 5
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/56/NCT05089656/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-28): https://cdn.clinicaltrials.gov/large-docs/56/NCT05089656/SAP_001.pdf